CLINICAL TRIAL: NCT02985918
Title: Effect of High-Intensity vs Low-Intensity Noninvasive Positive Pressure Ventilation on the Need for Endotracheal Intubation in Patients With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease The HAPPEN Randomized Clinical Trial
Brief Title: High-Intensity vs Low-Intensity NPPV in Patients With an AECOPD: The HAPPEN Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial has been terminated by the DSMB and the trial steering committee, based on the interim analysis results and the impracticality of continuing the trial in the context of the coronavirus disease 2019 (COVID-19) pandemic.
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, Principal Investigator, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeijingCYH-ICU-004
Record Dates: First submitted 2016-12-02; First posted 2016-12-07 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity NPPV (Experimental): Patients will receive high-intensity NPPV.
  Interventions: Device: High-intensity NPPV
- Low-intensity NPPV (Active Comparator): Patients will receive low-intensity NPPV.
  Interventions: Device: Low-intensity NPPV

INTERVENTIONS:
Device: High-intensity NPPV — In the high-intensity NPPV group, IPAP is initially adjusted in increments/decrements of 1-2 cmH2O, typically ranging from 20 to 30 cmH2O (or a tolerated maximum), to obtain a VT 10-15 mL/kg PBW and a respiratory rate <25 breaths/min. Subsequent adjustments to IPAP are based on the results of arterial blood gases (ABGs; up to 30 cmH2O) to achieve normocapnia (if possible), or to maximally decrease PaCO2 toward normocapnia if normocapnia can not be achieved. If PaCO2 decreases to less than 35 mmHg, IPAP will be decreased to achieve normocapnia.
  Arms: High-intensity NPPV
Device: Low-intensity NPPV — In the low-intensity NPPV group, as well as during the 6-hour trial of low-intensity NPPV, IPAP is initially adjusted in increments/decrements of 1-2 cmH2O (up to 20 cmH2O), according to patients' tolerance, to obtain a VT 6-10 mL/kg PBW and a respiratory rate <25 breaths/min. Subsequent adjustments to IPAP are based on the results of ABGs (up to 20 cmH2O) to achieve a pH of ≥7.35 and to reduce PaCO2 to a level deemed appropriate by the attending physician.
  Arms: Low-intensity NPPV

SUMMARY:
To determine whether high-intensity NPPV, compared with low-intensity NPPV, could reduce the need for endotracheal intubation during hospitalization in patients with an AECOPD and hypercapnia.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD confirmed by the 2019 criteria of the Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* Arterial pH <7.35 and PaCO2 >45 mmHg at screening entry
* PaCO2 >45 mmHg after a 6-hour trial of low-intensity NPPV

Exclusion Criteria:

* Age <18 years
* Excessive respiratory secretions with weak cough
* Upper airway obstruction
* Recent oral, facial, or cranial trauma or surgery
* Recent gastric or esophageal surgery
* Presence of restrictive ventilatory dysfunction (eg, consolidation or removal of at least one pulmonary lobe, massive pleural effusion, chest wall deformity, continuous strapping with thoracic or abdominal bandage, or severe abdominal distension)
* Active upper gastrointestinal bleeding
* Cardiac or respiratory arrest
* Arterial oxygen tension/fraction of inspired oxygen (PaO2/FiO2) <100 mmHg
* Pneumothorax
* Obvious emphysematous bullae confirmed by chest CT scan
* Ventricular arrhythmia or myocardial ischemia
* Severe hemodynamic instability (mean arterial pressure <65 mmHg)
* Severe metabolic acidosis (pH <7.20 and bicarbonate <22 mmol/L)
* Refusal to receive NPPV or give informed consent
* Prior endotracheal intubation or tracheostomy during the current hospitalization
* A do-not-intubate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
The need for endotracheal intubation during hospitalization | From randomization to discharge from hospital
  Defined as the proportion of patients who needed for endotracheal intubation during hospitalization after randomization

SECONDARY OUTCOMES:
Actual intubation during hospitalization | From randomization to discharge from hospital
  Defined as the proportion of patients actually receiving intubation and invasive ventilation during hospitalization after randomization
Need for endotracheal intubation at day 28 | Within 28 days since randomization
  Defined as the proportion of patients who needed endotracheal intubation within 28 days since randomization
Actual intubation at day 28 | Within 28 days since randomization
  Defined as the proportion of patients receiving intubation and invasive ventilation within 28 days after randomization
The composite of actual intubation or avoiding intubation by crossover to high-intensity NPPV | From randomization to discharge from hospital
  Defined as the incidence of patients receiving actual intubation in the high-intensity NPPV group vs the composite incidence of actual intubation or avoiding intubation by crossover to high-intensity NPPV in case of intubation criteria in the low-intensity NPPV group) during hospitalization after randomization
NPPV weaning success | From randomization to discharge from hospital
  Defined as the proportion of patients with persistent disconnection of NPPV without the presence of respiratory distress within the following 72 hours during hospitalization after randomization
Mortality in hospital | From randomization to discharge from hospital
Mortality at day 28 | Within 28 days since randomization
Mortality at day 90 | Within 90 days since randomization
Intensive care unit admission | From randomization to discharge from hospital
  Defined as the proportion of patients who transferred to ICU during hospitalization after randomization
Live discharge from the hospital | From randomization to discharge from hospital
  Defined as the proportion of patients with the exception of those who died and withdrawn treatment therapy during hospitalization after randomization.
Length of hospital stay | From hospital admission to discharge
  Defined as the number of days for the index hospitalization
Length of hospital stay after randomization | From randomization to discharge from hospital
  Defined as the number of hospitalization days since randomization
Invasive ventilator-free days at day 28 | Within 28 days since randomization
  Defined as 28 minus the number of days with invasive ventilator (range, 0-28 days) since randomization
ICU-free days at day 28 | Within 28 days since randomization
  Defined as 28 minus the number of days in the ICU (range, 0-28 days) since randomization
Hospital readmission at day 90 | Within 90 days since randomization
  Defined as the number of hospitalization days within 90 days since randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zujin Luo, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (31):
- China (31):
  - Wuyuan Hospital of Inner Mongolia, Bayan Nur
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Fangshan Liangxiang Hospital,, Beijing
  - Beijing Jingmei Group General Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Beijing Mentougou District Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Beijing Zhongguancun Hospital, Beijing
  - Capital Medical University Daxing Teaching Hospital, Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Dalian Friendship Hospital, Dalian
  - Dalian Municipal Central Hospital, Dalian
  - Shulan (Hang Zhou) Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Hemei General Hospital, Hebi
  - Huangshi Central Hospital, Huangshi
  - Jiaozuo People's Hospital, Jiaozuo
  - Jiaozuo Second Hospital, Jiaozuo
  - Kaifeng Central Hospital, Kaifeng
  - The First Affiliated Hospital of Hanan University,, Kaifeng
  - The First People's Hospital of Luoyang, Luoyang
  - The Third Hospital of Mianyang, Mianyang
  - Nanyang Central Hospital, Nanyang
  - Nanyang First People's Hospital, Nanyang
  - Sanmenxia Central Hospital, Sanmenxia
  - The Second Hospital of Tongliao, Tongliao
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi
  - Xinxiang Central Hospital, Xinxiang
  - Zhengzhou Central Hospital, Zhengzhou
  - Hunan Province Directly Affiliated TCM Hospital, Zhuzhou
  - Zibo First Hospital, Zibo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Z, Li Y, Li W, Li Y, Nie Q, Shi Y, Wang J, Ji Q, Han X, Liu S, Li D, Wang S, Li Z, Jia D, Ge H, Xu P, Feng Z, Li F, An F, Tai N, Yue L, Xie H, Jin X, Liu H, Dang Q, Zhang Y, Sun L, Wang J, Huang H, Chen L, Ma Y, Cao Z, Wang C; HAPPEN Investigators. Effect of High-Intensity vs Low-Intensity Noninvasive Positive Pressure Ventilation on the Need for Endotracheal Intubation in Patients With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease: The HAPPEN Randomized Clinical Trial. JAMA. 2024 Nov 26;332(20):1709-1722. doi: 10.1001/jama.2024.15815. PMID 39283649
- [Derived] Luo Z, Wu C, Li Q, Zhu J, Pang B, Shi Y, Ma Y, Cao Z; HAPPEN collaboration group. High-intensity versus low-intensity noninvasive positive pressure ventilation in patients with acute exacerbation of chronic obstructive pulmonary disease (HAPPEN): study protocol for a multicenter randomized controlled trial. Trials. 2018 Nov 21;19(1):645. doi: 10.1186/s13063-018-2991-y. PMID 30463622